CLINICAL TRIAL: NCT04298060
Title: A Phase IIb Randomized Placebo-Controlled Study to Examine the Efficacy and Safety of DAS181 for the Treatment of Severe Influenza Infection
Brief Title: DAS181 for Patients With Severe Hospitalized Flu and SAD-RVs (COVID-19)
Acronym: STOP-Flu
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ansun Biopharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DAS181-2-07
Record Dates: First submitted 2020-02-28; First posted 2020-03-06 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Influenza Infection; SAD-RV Infection and COVID-19
Keywords: Severe hospitalized influenza; Lower Respiratory Tract Disease; Acute Hypoxemia; DAS181; Ansun; infection
MeSH Terms: conditions — COVID-19; Infections | interventions — oplunofusp

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Stage 2, Ansun will know the dosage.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- DAS181 SD group Cohort 1, Stage 1 (Experimental): DAS181 SD group 4.5mg/day for 7 or 10 days
  Interventions: Drug: DAS181
- DAS181 HD group Cohort 1, Stage 1 (Experimental): DAS181 HD group 9mg/day for 7 or 10 days.
  Interventions: Drug: DAS181
- Placebo, Cohort 1, Stage 1 (Placebo Comparator): Placebo 0mg/day for 7 or 10 days
  Interventions: Drug: Placebo
- DAS181 group, Cohort 1, Stage 2 (Experimental): DAS181 4.5mg/day or 9mg/day. Dosage will be determined after completion of stage 1.
  Interventions: Drug: DAS181
- Placebo, Cohort 1, Stage 2 (Placebo Comparator): Placebo 0mg/day for 7 or 10 days
  Interventions: Drug: Placebo
- DAS181 group, Cohort 2, Stage1 and 2 (Experimental): DAS181 4.5mg/day or 9mg/day for 7 or 10 days
  Interventions: Drug: DAS181

INTERVENTIONS:
Drug: DAS181 — SD (4.5mg/day), HD (9mg/day)
  Arms: DAS181 HD group Cohort 1, Stage 1; DAS181 SD group Cohort 1, Stage 1; DAS181 group, Cohort 1, Stage 2; DAS181 group, Cohort 2, Stage1 and 2
Drug: Placebo — Placebo 0mg/day
  Arms: Placebo, Cohort 1, Stage 1; Placebo, Cohort 1, Stage 2

SUMMARY:
This is a Phase IIb study consisting of two cohorts to evaluate efficacy, safety and pharmacokinetics of DAS181 in IFV infection. An approximate total of 280 subjects will be enrolled into this study.

DETAILED DESCRIPTION:
Cohort 1: It is designed as a two stage, multi-center, randomized, double-blind, two parallel doses, placebo-controlled study that will investigate the efficacy of DAS181 for the treatment of serious IFV in hospitalized patients who suffered from acute hypoxemia requiring supplemental oxygen therapy.

Cohort 2: It is designed as an open-label study that will investigate the efficacy of DAS181 for the treatment of patients with sever IFV but not eligible for Cohort 1 and non-IFV SAD viral infection, e.g. parainfluenza virus, human metapneumovirus, enterovirus and all strains of β-coronaviruses (including but not limited to SARS-CoV-2), with hypoxemia requiring supplemental oxygen therapy.

ELIGIBILITY:
Inclusion criteria of Cohort 1 #4 is adapted from the Flu guideline in China (2018) and community acquired pneumonia (CAP) guideline in China (2016)

Cohort 1:

Subjects must meet all of the following inclusion criteria at the time of randomization to be eligible for participation in this study:

1. Males and Females ≥18 years old
2. Diagnosed as influenza (IFV) infection within 3 days before randomization
3. Requires, at the time of randomization, supplemental oxygen ≥2 LPM due to hypoxemia
4. Subjects are severely ill
5. In the opinion of investigator, subjects will be hospitalized at least 1 week.
6. If female, subject must not be pregnant or nursing

Cohort 2:

Subjects must meet all of the following inclusion criteria at the time of randomization to be eligible for participation in this study:

1. Males and Females ≥18 years old
2. Hypoxemia
3. Subjects fulfill one of the following conditions:

   1. IFV subjects who are eligible for all inclusion criteria of Cohort 1 except for acute hypoxemia at enrollment.
   2. Subjects confirmed with non-IFV SAD viral infection.
4. Same in inclusion criteria #5 to #8 in Cohort 1.

Exclusion Criteria

Cohort 1 and 2:

Subjects who meet any of the following exclusion criteria are not to be enrolled in this study:

1. Subjects requiring mechanical, Bi-PAP or CPAP ventilation at randomization.
2. Life expectancy less than 30 days.
3. Subjects with conscious disturbance (slow response, drowsy, restlessness, anxiety, confusion, twitching or convulsion)
4. Subjects with unstable hemodynamics such as systolic blood pressure < 90 mmHg or septic shock
5. Subjects with BUN≧7.14 mmol/L
6. Subjects treated with inhaled anti-viral therapy and washout period ≦ 48 hours.
7. If Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST) or Alkaline Phosphatase (ALP) are ≥3x ULN and Total Bilirubin (TB) is ≥2x ULN.
8. Female subjects with positive pregnancy test result, breastfeeding or planning to breastfeed at any time through 30 days after the last dose of study drug.
9. Subjects taking any other investigational drug used to treat for another respiratory infection.
10. Psychiatric or cognitive illness or recreational drug/alcohol use that, in the opinion of the principal investigator, would affect subject safety and/or compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2020-07 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Percent of subjects who have returned to room air | 7 days
  Percent of subjects who have returned to room air
Percent change of subjects return to baseline oxygen requirement | 7 days
  Percent change of subjects return to baseline oxygen requirement by Day 7 compared to Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Ho, MD, PhD, Study Director — Ansun Biopharma, Inc.
Locations (1):
- Ruijin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, China